CLINICAL TRIAL: NCT03024372
Title: A Prospective Randomized Single Blinded Study of Continuous Suturing Versus Interrupted Clips for Brachiocephalic AV Fistula Creation
Brief Title: Continuous Suturing Versus Interrupted Clips for Brachiocephalic AV Fistula Creation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not get started. Investigator is no longer at this institution
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sutures vs Clips AVF
Record Dates: First submitted 2017-01-06; First posted 2017-01-18 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2017-10

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Sutures; Surgical Instruments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional sutures (Active Comparator): AV fistula creation with sutures
  Interventions: Device: AV Fistula creation with sutures
- Anastoclips (Active Comparator): AV fistula creation with clips
  Interventions: Device: AV Fistula creation with clips

INTERVENTIONS:
Device: AV Fistula creation with sutures — End-to-side anastomosis (of AV fistula) is to be constructed using sutures. The incision is to be irrigated and closed using Vicryl, Biosyn and skin glue.
  Arms: Conventional sutures
Device: AV Fistula creation with clips — End-to-side anastomosis (of AV fistula) is to be constructed using clips. The incision is to be irrigated and closed using Vicryl, Biosyn and skin glue.
  Arms: Anastoclips

SUMMARY:
The purpose of this study is to investigate a promising strategy to improve maturation and patency rates following creation of AV fistulas and assess whether an anastomosis performed with Anastoclips (interrupted, nonpenetrating) would produce better maturation and/or patency than one performed with conventional suturing techniques.

DETAILED DESCRIPTION:
This will be a single blind (patient and dialysis center), prospective, randomized trial conducted at a single center. The study intervention will be randomization between conventional sutured anastomosis (Control group) and use of Anastoclips (Treatment group), which provide an interrupted closure without intimal penetration.

ELIGIBILITY:
Inclusion Criteria:

* Requiring brachiocephalic fistula judged to be best option for access after vein mapping (Surgeons will be required to do 10 cases using Anastoclips prior to enrolling)
* Able to provide informed consent in English or Spanish
* Age 18 years or greater
* With estimated life expectancy of 2 years or more
* Able to comply with study procedures including all scheduled follow-up visits

Exclusion Criteria:

* Unable to provide informed consent in English or Spanish
* Age < 18 years
* With pacemaker, IACD, or other permanent obstructive device on that side (a temporary tunneled dialysis catheter is not an exclusion)
* Unable (or in surgeon's judgment a poor risk) to comply with study procedures and follow-up visits
* With estimated life expectancy of less than 2 years
* Females must be either:

  * Of non-childbearing potential, which is defined as post-menopausal (at least 12 months without menses prior to Treatment Day) or documented surgically sterile or post hysterectomy (at least 1 month prior to Treatment Day)
  * Or, of childbearing potential, in which case must have a negative urine pregnancy test at Treatment Day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Time to loss of primary patency | one year post surgery

SECONDARY OUTCOMES:
Time to loss of secondary patency | one year post surgery
Time to loss of assisted primary patency | one year post surgery
Rate of functional maturation | one year post surgery
  in patients on dialysis
Time to functional maturation | one year post surgery
  in patients on dialysis
Rate of assumed maturation | one year post surgery
  in patients not on dialysis
Time to assumed maturation | one year post surgery
  in patients not on dialysis
Rate of complications | 30 days post surgery
  thrombosis/thrombectomy, stenosis, skin erosion, limb swelling, steal syndrome, bleeding and hematoma formation at surgical site, surgical-site-related infection, access-related infection, rupture, revision
Rate of intervention | five years post surgery
  to maintain patency
Operative cost | duration of surgery
Overall cost | time of surgery to time of hospital discharge (can range from 1 day to 1 week or more)
  Overall cost of surgery itself defined as from surgery to point of hospital discharge, anticipated to be in days
Time to loss of primary patency | 5 years post surgery
Time to loss of assisted primary patency | 5 years post surgery
Time to loss of secondary patency | 5 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karl Illig, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida - South Tampa Campus, Tampa, Florida
  - USF Health Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haruguchi H, Nakagawa Y, Uchida Y, Sageshima J, Fuchinoue S, Agishi T. Clinical application of vascular closure staple clips for blood access surgery. ASAIO J. 1998 Sep-Oct;44(5):M562-4. doi: 10.1097/00002480-199809000-00050. PMID 9804495
- [Background] Schild AF, Pruett CS, Newman MI, Raines J, Petersen F, Konkin T, Kim P, Dickson C, Kirsch WM. The utility of the VCS clip for creation of vascular access for hemodialysis: long-term results and intraoperative benefits. Cardiovasc Surg. 2001 Dec;9(6):526-30. doi: 10.1016/s0967-2109(01)00088-6. PMID 11604333
- [Background] Cook JW, Schuman ES, Standage BA, Heinl P. Patency and flow characteristics using stapled vascular anastomoses in dialysis grafts. Am J Surg. 2001 Jan;181(1):24-7. doi: 10.1016/s0002-9610(00)00547-x. PMID 11248171
- [Background] Cooper BZ, Flores L, Ramirez JA, Najjar JG, Abir F, Rayham R, Paladino L, Nguyen M, Panetta TF. Analysis of nonpenetrating clips versus sutures for arterial venous graft anastomosis. Ann Vasc Surg. 2001 Jan;15(1):7-12. doi: 10.1007/s100160010001. PMID 11221948
- [Background] Zeebregts CJ. Randomized clinical trial of continuous sutures or non-penetrating clips for radiocephalic arteriovenous fistula (Br J Surg 2004; 91: 1438-1442). Br J Surg. 2005 May;92(5):654-5. doi: 10.1002/bjs.5063. No abstract available. PMID 15852413
- [Background] Sukhatme VP. Vascular access stenosis: prospects for prevention and therapy. Kidney Int. 1996 Apr;49(4):1161-74. doi: 10.1038/ki.1996.167. No abstract available. PMID 8691738
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Sidawy AN, Gray R, Besarab A, Henry M, Ascher E, Silva M Jr, Miller A, Scher L, Trerotola S, Gregory RT, Rutherford RB, Kent KC. Recommended standards for reports dealing with arteriovenous hemodialysis accesses. J Vasc Surg. 2002 Mar;35(3):603-10. doi: 10.1067/mva.2002.122025. PMID 11877717
- [Background] Zhou XH, Melfi CA, Hui SL. Methods for comparison of cost data. Ann Intern Med. 1997 Oct 15;127(8 Pt 2):752-6. doi: 10.7326/0003-4819-127-8_part_2-199710151-00063. PMID 9382393
- [Result] Shenoy S, Miller A, Petersen F, Kirsch WM, Konkin T, Kim P, Dickson C, Schild AF, Stewart L, Reyes M, Anton L, Woodward RS. A multicenter study of permanent hemodialysis access patency: beneficial effect of clipped vascular anastomotic technique. J Vasc Surg. 2003 Aug;38(2):229-35. doi: 10.1016/s0741-5214(03)00412-9. PMID 12891102
- [Result] Nguyen KP, Teruya T, Alabi O, Sheng N, Bianchi C, Chiriano J, Dehom S, Abou-Zamzam A. Comparison of Nonpenetrating Titanium Clips versus Continuous Polypropylene Suture in Dialysis Access Creation. Ann Vasc Surg. 2016 Apr;32:15-9. doi: 10.1016/j.avsg.2015.11.008. Epub 2016 Jan 22. PMID 26806237
- [Result] Aitken E, Jeans E, Aitken M, Kingsmore D. A randomized controlled trial of interrupted versus continuous suturing techniques for radiocephalic fistulas. J Vasc Surg. 2015 Dec;62(6):1575-82. doi: 10.1016/j.jvs.2015.07.083. Epub 2015 Oct 23. PMID 26506936
- [Result] Zeebregts C, van den Dungen J, Buikema H, van der Want J, van Schilfgaarde R. Preservation of endothelial integrity and function in experimental vascular anastomosis with non-penetrating clips. Br J Surg. 2001 Sep;88(9):1201-8. doi: 10.1046/j.0007-1323.2001.01857.x. PMID 11531868